CLINICAL TRIAL: NCT01203865
Title: Prevalence of Fibromyalgia in Israel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0303-10-TLV; WS573984 (Other Grant/Funding Number: Pfizer Inc.)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Fatigue
MeSH Terms: conditions — Fibromyalgia; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of fibromyalgia syndrome in the Israeli population is of importance fro planning resource allocation of medical expenditure as well as for identifying demographic and ethnic differences of this unique population compared with other western samples. In the current study the investigators aim at estimating the prevalence of fibromyalgia in this population. For this purpose a two - stage process will be used. First, a population survey will be conducted by telephone, screening for widespread pain and fatigue in the general population. This survey will use the London Fibromyalgia Epidemiology Study Screening Questionnaire. Second, a sample of patients attending the rheumatology clinic will be surveyed with this tool and will be examined in order to determine the actual proportion of patients fulfilling ACR criteria for fibromyalgia. This will enable us to calculate the positive predictive value of the London Fibromyalgia Epidemiology Study Screening Questionnaire in our population and hence to calculate the prevalence of fibromyalgia in the population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 who consent to answer the survey questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Telephone survey - general population over age 18 Rheumatology patients - patients attending the rheumatology clinic for any reason
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-11 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of fibromyalgia in the Israeli population | 9 months

SECONDARY OUTCOMES:
Demographic data on fibromyalgia patients | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacob N Ablin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv SOurasky Medical center, Tel Aviv, Israel

REFERENCES:
- [Background] Branco JC, Bannwarth B, Failde I, Abello Carbonell J, Blotman F, Spaeth M, Saraiva F, Nacci F, Thomas E, Caubere JP, Le Lay K, Taieb C, Matucci-Cerinic M. Prevalence of fibromyalgia: a survey in five European countries. Semin Arthritis Rheum. 2010 Jun;39(6):448-53. doi: 10.1016/j.semarthrit.2008.12.003. Epub 2009 Feb 27. PMID 19250656